CLINICAL TRIAL: NCT06148142
Title: Effectiveness of a Community Pharmacy-based Health Promotion Program on Hypertension in Bangladesh and Pakistan: Study Protocol for a Cluster Randomized Controlled Trial
Brief Title: Effectiveness of a Community Pharmacy-based Health Promotion Program on Hypertension in Bangladesh and Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitotsubashi University (Other)
Collaborators: Global Public Health Research Foundation (Other)
Responsible Party: Principal Investigator, Md. Mizanur Rahman, PhD, Associate Professor, Hitotsubashi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023D016
Record Dates: First submitted 2023-11-07; First posted 2023-11-28 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Blood Pressure; Pharmacy; Cost-effectiveness
Keywords: Hypertension control; quality-adjusted life year gained; Cost-effectiveness; South Asia

STUDY DESIGN:
Intervention Model Description: Two-arm cluster randomized controlled trial (cRCT) will be conducted among hypertensive subjects in Bangladesh and Pakistan.
Who Masked: Participant
Masking Description: Only the outcome evaluators will be blinded from group allocation due to the nature of the intervention. CP will deliver the intervention and research assistants (field enumerators and supervisors) will engage in data collection from the participants. However, pharmacists and research assistants will not be blinded since they are involved in interventional processes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assigned Interventions (Experimental): The intervention to experimental/intervention group will consist of three phases: baseline survey with first time intervention implementation; second intervention at 6 months; third at 12 months and , end-line survey at 18 months. As part of the intervention within the randomized selected groups, the CP will conduct two 15-30 minute sessions throughout the intervention period, once at the baseline or first visit (T0) and once at the sixth month (T1). Face-to-face counselling sessions will be held about hypertension and its management, including lifestyle changes and drug compliance. Patients will be able to view the educational material in the pharmacy via a tablet, since audio-visual presentations make learning easier. The intervention group will receive phone call intervention at 3 months and 6 months.
  Interventions: Behavioral: Pharmacy based health promotion
- Control group (Active Comparator): In the control group, routine pharmacy services and counselling will be provided without interference during all-pharmacy visits, as per each country's pharmacy practice guidelines, and they will serve as a comparator group to determine the impact of the intervention implementation. Assessments will be completed at the same time points as those in the intervention group.
  Interventions: Behavioral: Pharmacy based health promotion

INTERVENTIONS:
Behavioral: Pharmacy based health promotion — This project will consist of three phases: baseline survey with first time intervention implementation; second intervention at 6 months; third at 12 months and , end-line survey at 18 months. As part of the intervention within the randomized selected groups, the CP will conduct two 15-30 minute sessions throughout the intervention period, once at the baseline or first visit (T0) and once at the sixth month (T1). Patients will attend the two sessions at the pharmacies where they collect their prescription medication. Face-to-face counselling sessions will be held about hypertension and its management, including lifestyle changes and drug compliance.

SUMMARY:
The aim of this multi-country research project is to reduce the blood pressure of individuals with hypertension over a 18-month period in Bangladesh and Pakistan. A cluster randomized controlled trial (cRCT) will be conducted with two arms. The estimated sample size is around 3600 hypertensive adults. Bangladesh study participants will consist of 3600 hypertensive individuals. Approximately 10% of participants will be selected based on Bangladesh samples from Pakistan (360 hypertensive patients, four pharmacies). Community pharmacies will be randomised to one of two parallel groups (allocation ratio 1:1). Pharmacy professionals will provide educational training and counselling, as well as phone calls/mobile text messages and care coordination in the health sector as part of the intervention. The study will be conducted in three phases: baseline survey; intervention and follow-up; and endline survey with impact evaluation. The primary outcome will be BP reduction and the secondary outcomes will be BP controlled to target, treatment adherence, mortality or hospital admission rates resulting from hypertension and its related complications, incremental cost per quality-adjusted life year gained, improvement in knowledge on healthy lifestyle, change in dietary salt intake, and change in prevalence of current smokers.

DETAILED DESCRIPTION:
Globally, hypertension is a leading cause of cardiovascular disease and death. Approximately two-thirds of the world's 1.28 billion hypertensive adults live in low- and middle-income countries (LMICs). South Asian countries have experienced a steep rise in hypertension prevalence, with Bangladesh, India, and Pakistan having 48.0%, 52.3%, and 46.2%. Hypertension in low-income countries is disproportionately caused by rapid urbanization, unhealthy lifestyles, and inactivity. In LMICs, though awareness, treatment, and control of hypertension remain unacceptably low, mostly because of poor medication adherence, limited health resources, and difficulties accessing healthcare. Furthermore, a systematic review suggested that factors such as inadequate health care information, dissatisfaction with the services provided, and fewer interactions with physicians contribute significantly to medication nonadherence. LMICs with weak health literacy, poor health systems, and high cardiovascular disease fatality rates have a disproportionately high prevalence of hypertension. Consequently, most hypertensive individuals take medications only when symptomatic and lead sedentary lifestyles despite being aware of dietary recommendations. Therefore, this study aims to evaluate the impact and cost-effectiveness of enhanced pharmacist care on blood pressure (BP) control and treatment adherence across two South Asian countries.

Objectives:

In this study, the investigator will test the effectiveness and cost-effectiveness of enhanced pharmacy-based care provided to community people in two South Asian countries (Bangladesh and Pakistan) on blood pressure control and treatment adherence. It is the first multi-country trial to evaluate pharmacy-based health promotion in these two countries, focusing on the role of pharmacist in hypertension treatment. This study hypothesizes that hypertensive participants receiving the community pharmacy-based health intervention will achieve the following:

* Reduced SBP and/or DBP;
* Treatment adherence and BP controlled to target (SBP 140 mmHg and DBP 90 mmHg) increased;
* Cardiovascular disease, heart failure or stroke are less likely to cause hospitalizations.
* Hypertension management costs are reduced;
* Changes in lifestyle behaviors, such as reducing salt intake, smoking, and physically inactivity.

Methods:

Study design and setting:

Two-arm cluster randomized controlled trial (cRCT) will be conducted among hypertensive subjects in Bangladesh and Pakistan. Randomization clusters are community pharmacies. Each country will follow a two-arm cRCT design. According to 4.65% BP reduction with 49.78 standard deviation, the estimated sample size for Bangladesh is around 3600 at 80% power and 5% significance. Approximately 10% of participants will be selected based on Bangladesh sample from Pakistan (360 hypertensive patients, four pharmacies). The average number of hypertensive participants per pharmacy is 90.

Study participants:

As part of the census, participants who come to the pharmacy to purchase hypertensive medication will be listed with their basic information. The following information will be needed: their name, address, gender, duration of hypertension, who will be taking the medication, and at least two contact numbers. In order to confirm whether prospective hypertensive participants are hypertensive, their blood pressure will be measured again. Both male and female participants will be invited to participate. The eligibility criteria include: (1) aged 18 years and above, (2) hypertensive (defined (a) SBP ≥140 mmHg and DBP ≥90 mmHg and/or taking antihypertensive medications), (3) having suboptimal medication adherence to antihypertensive drugs according to the Morisky Medication Adherence Scale, (4) capable of communicating verbally in local language, (5) permanent resident of the study area, (6) access to mobile phone, and (7) consent to participate. Exclusion criteria will be: (1) pregnant and lactating women, (2) individuals with advanced medical disease, (3) those having cognitive and psychiatric problems, (4) involvement in any other interventional study, and (5) individuals who are unable to give informed consent. Pharmacists' inclusion criteria include: (1) ensuring sufficient amount of time to implement intervention on hypertensive participants, (2) consent to participate and (3) able to operate smartphone or tablet. Screening for patients' eligibility will be conducted by the CP during regular visits, and upon deeming them eligible, the CP will inform the principal investigator or research assistant of this study to approach the patients, briefly explain the study, and ask to sign informed consent.

Randomization: Community pharmacies will then be randomised to one of two parallel groups (allocation ratio 1:1) using a computer-generated random number sequence. Participants and pharmacies will be assigned to intervention and control groups in a 1:1 ratio.

Training of the pharmacists:

A mandatory communication training will enhance treatment integrity, since pharmacist skills and competences will determine the quality of the intervention. Before the study begins, CP in the intervention arm will receive a training involving both theoretical and practical sessions. It will cover prevalence, risk factors, complications, and diagnosis of hypertension, as well as non-pharmacological ways of preventing it. On the practical side, CPs will learn how to measure blood pressure using a manual sphygmomanometer, interpret the measurements, and educate and counsel hypertensive patients through audio-visual presentations. As part of the intervention strategy, blood pressure control, identification of hypertension-related complications, health education, medication and lifestyle modification counselling, follow-up, and referral to a medical practitioner or hospital will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years to 90 years old
* Hypertensive (SBP ≥140 mmHg and DBP ≥90 mmHg and/or taking antihypertensive medications)
* Having suboptimal medication adherence to antihypertensive drugs
* Capable of communicating verbally in local language
* Permanent resident of the study area
* Access to mobile phone
* Consent to participate

Pharmacists' inclusion criteria include:

* Ensuring a sufficient amount of time to implement intervention on hypertensive participants
* Consent to participate
* Able to operate smartphone or tablet.

Exclusion Criteria:

* Pregnant and lactating women
* Individuals with advanced medical disease
* Those having cognitive and psychiatric problems,
* Involvement in any other interventional study
* Individuals who are unable to give informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3600 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure change | Participants will be assessed at baseline, at baseline, at 12 months and 18 months post-intervention
  The primary effectiveness of the outcome will be evaluated by change in SBP and DBP of the patients at baseline, at 12 months and 18 months post-intervention.

SECONDARY OUTCOMES:
Changes in blood pressure from baseline to follow up | Participants will be assessed at baseline, at baseline, at 12 months and 18 months post-intervention
  Changes in Blood pressure in the target intervention group (Whose SBP<140 mmHg and DBP<90 mmHg were in the baseline)
Changes of Quality of life | Participants will be assessed at baseline, at baseline, at 12 months and 18 months post-intervention
  The incremental cost per quality-adjusted life year (QALY) gained from baseline to end of follow-up.
Knowledge of healthy lifestyle | Participants will be assessed at baseline, at baseline, at 12 months and 18 months post-intervention
  Improvement in the knowledge of patients on healthy lifestyle measurement by questionnaire.
Changes in salt intake | Participants will be assessed at baseline, at baseline, at 12 months and 18 months post-intervention
  Change in dietary salt intake by questionnaire.
Rate of treatment adherence | Time Frame: Participants will be assessed at baseline, at baseline, at 12 months and 18 months post-intervention
  Adherence to treatment adherence by questionnaires and hypertensive drug adherence by Morisky Medication Adherence Scale (MMAS-8)

CONTACTS AND LOCATIONS:
Locations (1):
- Global Public Health Research Foundation, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No